CLINICAL TRIAL: NCT04525443
Title: Assessment of Endothelial Vasodilator Function in COVID-19 Patients
Brief Title: Endothelial Function and COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hernan D. Mejia-Renteria, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: 20/451
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: Endothelial function; Endothelial cells; Blood vessels
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with active SARS-CoV-2 infection.: Patients admitted for COVID-19 at Hospital Clínico San Carlos with positive SARS-CoV-2 polymerase chain reaction (PCR).
- Patients with past, not active, SARS-CoV-2 infection.: Patients with past infection (not active), demonstrated by serology and PCR.
- People without concurrent or past SARS-CoV-2 infection: Health personnel from the Cardiology Service of Hospital Clínico San Carlos who demonstrate by serology that they have not had SARS-CoV-2 infection.

SUMMARY:
The present study aims to investigate the endothelial vasodilator function in patients with COVID-19

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), secondary to infection by severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) has caused a global pandemic with significant adverse effects on the health, social and economic systems in different countries of the world.

The entry receptor utilized by SARS-CoV-2 is Angiotensin-Converting Enzyme 2 (ACE-2), localized at the membrane of epithelial and endothelial cells and muscle cells of blood vessels. Hypothetically, this interaction of SARS-CoV-2 with essential elements of the blood vessels may conduct to endothelial dysfunction. In fact, it has been demonstrated several degrees of endothelial compromise in the kidney, small bowel and lungs from histological analysis in fatidic cases.

The pathophysiological mechanisms by which vascular endothelial dysfunction can complicate the evolutionary course of viral infections are of two types:

1. On the one hand, acute endothelial dysfunction can produce ischemic events as a consequence of thrombotic or vasomotor processes. Some of these events are acute coronary syndromes, pulmonary thromboembolism and peripheral angiopathy, all of which have been reported in COVID-19 patients.
2. On the other hand, vascular endothelial dysfunction can trigger or amplify systemic inflammatory reactions leading to multi-organ failure. Vascular hyperpermeability generated by vascular endothelial dysfunction is key in the processes of infiltration of immune cells and in the amplification of the inflammatory response that occurs in the context of the cytokine storm associated with the viral infection. This process contributes to release large amounts of IL 6, IL-1B and TNF alpha by vascular endothelial cells, thus the expression of vascular adhesion molecules.

In this study, the investigators sought to evaluate the status of vascular endothelial function in COVID-19 patients from a non-invasive approach.

The evaluation of systemic vascular endothelial function will be performed non-invasively using peripheral arterial tonometry with EndoPat system (Itamar). It is a technique that determines the endothelial-dependent changes in arterial tone of the vascular network of the index finger of both hands. Using bio-sensors placed on the pad of the index finger of both hands, an assessment of arterial tone is carried out at three stages: 1) at baseline; 2) during an ischemia caused by the inflation of a pressure cuff in one of the arms to occlude the brachial artery for 5 minutes; 3) and in a situation of reactive hyperemia during the recovery of arterial irrigation after deflating the pressure cuff. The arterial tone signals detected by plethysmography at the three described times are converted into digital signals for each arm explored, and the EndoPat software automatically determines the hyperemic vascular response.

To avoid biases in the analysis of systemic vascular endothelial function in COVID-19 patients, the research team led by Dr. Amir Lerman from the Mayo Clinic, Rochester, USA will blindly carry out the analysis of the EndoPat results. For this, the EndoPat study reports will be sent in an analyzable format for each patient included in the study, completely anonymized and at blind fashion with respect to the group that patient belongs, the moment in which EndoPat assessment was made (days from the onset of symptoms in the case of the study group), blinded for the results of blood tests related to inflammation, and for the clinical evolution of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Study group No. 1: age ≥ 18 years; COVID-19 confirmed with positive PCR. Availability of informed consent.
* Study group No. 2: age ≥ 18 years; Past SARS-CoV-2 infection demonstrated by PCR and serology.
* Control group: age ≥ 18 years; absence of concurrent or previous SARS-CoV2 infection demonstrated by serology, and absence of acute or chronic diseases related to endothelial dysfunction, mainly acute or chronic infectious or inflammatory processes and known peripheral vascular disease.

Exclusion Criteria:

* Impossibility of performing the endothelial function test.
* Recent puncture of the radial artery (<15 days).
* Hemodynamic instability.
* Unavailability of signed informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population is made up of three group of patients:
  * Study group No. 1: patients with active SARS-CoV-2 infection.
  * Study group No. 2: patients with past, not active, SARS-CoV-2 infection.
  * Control group: People without concurrent or past SARS-CoV-2 infection. Group No. 1 will include patients admitted for COVID-19 at Hospital Clínico San Carlos with positive SARS-CoV-2 PCR; group 2 will include patients with past infection demonstrated by serology and PCR, and will be constituted by either health personnel from Hospital Clínico San Carlos who have passed the disease, or patients who have been discharged from the hospital; and the control group will include health personnel from the Cardiology Service of Hospital Clínico San Carlos who demonstrate by serology that they have not had SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Reactive hyperemia index (RHI) | Baseline
  RHI derived from peripheral arterial tonometry with EndoPat system (Itamar)

SECONDARY OUTCOMES:
Percentage of COVID-19 patients with impaired endothelial vasodilator function. | Up to 3 months
Percentage of non-COVID-19 patients with impaired endothelial vasodilator function. | Baseline

OTHER OUTCOMES:
Percentage variation of RHI during the evolutionary course of COVID-19. | At baseline and 1-3 months after COVID-19 resolution

CONTACTS AND LOCATIONS:
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Hospital Clínico San Carlos, Madrid, Spain